CLINICAL TRIAL: NCT01759485
Title: Vitamin D Supplementation as Adjunct to Clozapine-treated Chronic Schizophrenia Patients
Brief Title: Vitamin D for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geha Mental Health Center (Other)
Responsible Party: Principal Investigator, Amir Krivoy, Senior Psychiatrist, Geha Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMHC-VITD; 29-12 (Other: GMHC)
Record Dates: First submitted 2012-12-04; First posted 2013-01-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Clozapine Resistant Schizophrenia
Keywords: Clozapine; Schizophrenia; Vitamin-D; Treatment-resistant
MeSH Terms: conditions — Schizophrenia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Supplementation of Vitamin D as add-on to the regular anti-psychotic treatment
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Placebo as oral drops once weekly as add-on to the regular anti-psychotic treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin D3 — once weekly oral drops preparation at a daily dose of 2000 IU X 7 = 14,000 IU per week (about 60 drops each week).
  Other Names: Cholecalciferol
  Arms: Vitamin D
Drug: placebo
  Arms: Placebo

SUMMARY:
Background: Despite improvements in medications, treatment delivery and rehabilitation, schizophrenia outcomes remain suboptimal. There are a proportion of 30-40% treatment-resistant schizophrenia patients. Multiple lines of evidence suggest that vitamin D is a neuro-active steroid that acts on brain development, leading to alterations in brain neurochemistry and adult brain function. Early deficiencies have been linked with neuropsychiatric disorders, such as schizophrenia, and adult deficiencies have been associated with adverse brain outcomes, including Parkinson's disease, Alzheimer's disease, depression and cognitive decline. Ecological studies support a potential role for vitamin D in schizophrenia. These data include studies that have explored the association between schizophrenia and winter/spring birth and also the apparent increased incidence and prevalence of schizophrenia at higher latitudes. Objective: To evaluate the effect of vitamin-D supplementation on the mental state of clozapine-treated chronic schizophrenia patients, and the relation of disease severity to serum vitamin D levels. Methods: the investigators will use a prospective, interventional, longitudinal, double blinded, placebo-controlled, randomized design. The investigators will recruit 50 clozapine-treated chronic schizophrenia patients, with low level of serum vitamin-D, that will be randomly assigned (1:1 ratio) to receive either weekly oral drops of vitamin D (Cholecalciferol) or oral drops of placebo for 8 weeks follow-up. Repeated assessments will include: clinical severity scales (PANSS, CGI), side effects (SAS, BARS, clozapine side effects), cognitive (MoCA), metabolic parameters and laboratory data. Patients who were assigned to placebo will be supplemented with vitamin D after the 8 weeks period, and then will be assessed again with the same protocol of vitamin D treated patients. All participants will be assessed again after 24 weeks after vitamin D initiation. Analysis: the investigators will use on-way ANOVA with repeated measures for comparison of vitamin D and control groups. The investigators will apply intention to treat and LOCF.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age 18-65 years
3. Diagnosis of schizophrenia according to DSM-IV-TR criteria, as confirmed by two senior psychiatrists
4. Total PANSS score > 70
5. CGI-S > 3
6. Clozapine treatment for at least 18 weeks
7. Vitamin D deficiency: plasma 25-OH-Vitamin D <75 nmol/L (20-30 ng/mL)
8. Able to consume oral drops of vitamin-D
9. Able to sign informed consent

Exclusion Criteria:

1. Mental retardation
2. Organic brain disease
3. Known parathyroid disorder
4. Inborn/acquired vitamin D metabolism disorders
5. Patients already treated with vitamin D supplementation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale total score | Baseline to 8 weeks

SECONDARY OUTCOMES:
Change in the MoCA Cognitive composite score | Baseline to 8 weeks

OTHER OUTCOMES:
Change in Positive and Negative Syndrome Scale sub-scores | Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Geha Mental Health Center, Petah Tikva, Israel